CLINICAL TRIAL: NCT06435169
Title: Comparative Presence of Piriformis Syndrome in Patients With Lumbar Disc Bulging and Protrusion
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Other Study IDs: Yuzuncu Yil University Türkiye
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 38 patients with lumbar disc bulging: Lasegue's test, FAIR (Flexion Adduction Internal Rotation) test and, Freiberg's test will be performed in a single check-up for patients diagnosed with L4-L5 and/or L5-S1 Lumbar Disc Herniation (bulging) by lumbar Magnetic Resonance Imaging (MRI). The presence of Piriformis syndrome was investigated in these patients with Freiberg and FAIR tests.
  Interventions: Diagnostic Test: Lasegue's, Freiberg's and, FAIR (Flexion Adduction Internal Rotation) tests.
- 38 patients with lumbar disc protrusion: Lasegue's, FAIR (Flexion Adduction Internal Rotation) and, Freiberg's test will be performed in a single check-up for patients diagnosed with L4-L5 and/or L5-S1 Lumbar Disc Herniation (protrusion) by lumbar Magnetic Resonance Imaging (MRI). The presence of Piriformis syndrome was investigated in these patients with Freiberg and FAIR tests.
  Interventions: Diagnostic Test: Lasegue's, Freiberg's and, FAIR (Flexion Adduction Internal Rotation) tests.

INTERVENTIONS:
Diagnostic Test: Lasegue's, Freiberg's and, FAIR (Flexion Adduction Internal Rotation) tests. — The Straight Leg Raise test or Lasegue test, is also crucial in detecting disc herniation and neural compression. Lasègue's sign is said to be positive if the angle to which the leg can be raised (upon straight leg raising) before eliciting pain is <45°.The presence of Piriformis syndrome was investigated in these patients with Freiberg and FAIR tests. Freiberg's test elicits pain by passively internal rotation of the extended hip, when the patient is in supine. The purpose of this test is on the one hand stretching of the irritated Piriformis Muscle (PM), on the other hand provoking sciatic nerve compression. The FAIR test is a sensitive and specific test for detection if irritation of the sciatic nerve by the piriformis. FAIR stands for flexion, adduction and internal rotation. Also known as piriformis test.

SUMMARY:
Clinicians consider lumbar disc herniation more prominently in the differential diagnosis than piriformis syndrome, as it is the most common cause of sciatica, and this canalizes them to overlook that the sciatic nerve may be compressed by the piriformis muscle, below the L4-L5-S1 intervertebral disc levels.

As far as is known, there are no 'patient series' in the literature regarding the incidence of Piriformis syndrome in Lumbar Disc Herniation, only one case report has been found. This clinical study aims to reveal that Piriformis syndrome may also be present in patients with disc herniation on Magnetic Resonance Imaging (MRI), and that sometimes it may even be the main cause of sciatic nerve pain.

DETAILED DESCRIPTION:
In this study, the participants between the ages of 18-65, who were diagnosed with L4-L5 and/or L5-S1 Lumbar Disc Herniation (bulging and protrusion) by having a Lumbar MRI at the Faculty of Medicine Sports Medicine outpatient clinic, were reached through their contact numbers, and those who had not previously undergone waist/hip surgery and those who described unilateral sciatica complaints (hip-leg-foot pain and numbness) during the interview were invited to Yüzüncü Yıl University Faculty of Medicine Sports Medicine polyclinic and Lasegue's, Flexion Adduction Internal Rotation (FAIR) and Freiberg's tests were performed.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having unilateral sciatica
* Having disk herniation in the form of bulging or protrusion in a previous Lumbar Magnetic Resonance Imaging (MRI)

Exclusion Criteria:

* Having bilateral sciatica
* Having disc herniation in the form of extrusion or sequestration in a previous Lumbar Magnetic Resonance Imaging (MRI)
* Previous back and/or hip surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders between the ages of 18-65 with lumbar disc bulging or protrusion
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Lasegue's Test | Baseline
  The Straight Leg Raise test or Lasegue test, is also crucial in detecting disc herniation and neural compression. Lasègue's sign is said to be positive if the angle to which the leg can be raised (upon straight leg raising) before eliciting pain is <45°.
Freiberg's Test | Baseline
  Freiberg's test elicits pain by passively internal rotation of the extended hip, when the patient is in supine. The purpose of this test is on the one hand stretching of the irritated piriformis muscle, on the other hand provoking sciatic nerve compression.
FAIR (Flexion Adduction Internal Rotation) test | Baseline
  The FAIR test is a sensitive and specific test for detection if irritation of the sciatic nerve by the piriformis. FAIR stands for flexion, adduction and internal rotation. Also known as piriformis test.

CONTACTS AND LOCATIONS:
Locations (1):
- Volkan Şah, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No